CLINICAL TRIAL: NCT03080883
Title: A Phase III, Randomized, Controlled, Double-Blind Study Evaluating the Safety of Two Doses of Apixaban for Secondary Prevention of Cancer Related Venous Thrombosis in Subjects Who Have Completed at Least Six Months of Anticoagulation Therapy
Brief Title: Apixaban in Preventing Secondary Cancer Related Venous Thrombosis in Cancer Patients Who Have Completed Anticoagulation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACCRU-SC-1601; NCI-2017-00325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-SC-1601 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2017-03-10; First posted 2017-03-15 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Vein Thrombosis; Deep Vein Thrombosis; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Pulmonary Embolism; Splanchnic Vein Thrombosis
MeSH Terms: conditions — Intracranial Thrombosis; Venous Thrombosis; Hematologic Neoplasms; Neoplasm Metastasis; Pulmonary Embolism | interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (lower dose apixaban) (Experimental): Patients receive lower dose apixaban PO BID for 365 days.
  Interventions: Drug: Apixaban
- Group II (higher dose apixaban) (Experimental): Patients receive higher dose apixaban PO BID for 365 days.
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Given PO
  Other Names: BMS-562247; BMS-562247-01; Eliquis

SUMMARY:
This randomized phase III trial studies the best dose of apixaban and how well it works in preventing secondary cancer related venous thrombosis in cancer patients who have completed anticoagulation therapy. Apixaban may help in prevention by blocking some of the enzymes needed for venous thrombosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Any episode of major bleeding including fatal bleeding or clinically relevant non-major bleeding.

SECONDARY OBJECTIVES:

I. The proportion of patients who experienced at least one such bleeding event within 6 months of beginning treatment.

II. Venous thromboembolism (VTE) recurrence including deep vein thrombosis (DVT), pulmonary embolism (PE), fatal PE, or arterial thromboembolism.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive lower dose apixaban orally (PO) twice daily (BID) for 365 days.

GROUP II: Patients receive higher dose apixaban PO BID for 365 days.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute index (original venous thrombotic) event: lower extremity or upper extremity (jugular, innominate, subclavian, axillary, brachial) DVT, PE, splanchnic (hepatic, portal, splenic, mesenteric, renal, gonadal), or cerebral vein thrombosis for which the patient has received >= 180 days (but =< 365 days) of anticoagulant therapy prior to registration; the date, imaging modality, and location of index event will be required; the date of initiation and specific type of anticoagulants used will also be required
* Active cancer defined as metastatic disease and/or any evidence of cancer on cross-sectional or positron emission tomography (PET) imaging, cancer related surgery, chemotherapy or radiation therapy within the past 6 months; Note: non-melanoma skin cancer does not meet the cancer requirement
* Life expectancy >= 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
* Hemoglobin >= 8 g/dL obtained =< 30 days prior to registration
* Platelet count >= 50,000/mm^3 obtained =< 30 days prior to registration
* Alanine aminotransferase (ALT) or aspartate transaminase (AST) =< 3 x upper limit of normal (ULN) obtained =< 30 days prior to registration
* Calculated creatinine clearance must be >= 30 ml/min using the Cockcroft-Gault formula obtained =< 30 days prior to registration
* Negative serum or urine pregnancy test done =< 7 days prior to registration, for women of childbearing potential only;

  * Note: a woman of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal; menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes
* Ability to provide informed written consent
* Willing to undergo monthly follow-up assessment, either in person at the enrolling institution or by telephone

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

    * Note: women of child bearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 33 days after finishing the last dose
    * Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 93 days after finishing the last dose
    * Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements; however they must still undergo pregnancy testing as described in this section; note: investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy; investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception; highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly; at a minimum, subjects must agree to the use of one method of highly effective contraception as listed below:

      * Male condoms with spermicide
      * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena by WOCBP subject or male subject's WOCBP partner
      * Female partners of male subjects participating in the study may use hormone based contraceptives as one of the acceptable methods of contraception
      * IUDs, such as ParaGard
      * Tubal ligation
      * Vasectomy
      * Complete abstinence

        * Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs; acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence
* Active major bleeding
* Severe hypersensitivity reaction to apixaban (e.g., anaphylactic reactions)
* Current use of strong CYP3A4 inducers or inhibitors

  * NOTE: patients may be eligible if they transition to an alternative agent or are able to stop CYP3A4 inducer or inhibitor
* Current use of thienopyridine therapy (clopidogrel, prasugrel, or ticagrelor) that will be continued on study
* Severe liver disease (known cirrhosis Childs Pugh class B or C), or active hepatitis
* Documented venous thromboembolism while on therapeutic anticoagulation ("anticoagulation failure")
* Mechanical heart valve
* Documented hemorrhagic tendencies (e.g., hemophilia)
* Bacterial endocarditis
* Any of the following conditions:

  * Intracranial bleeding =< 6 months prior to randomization
  * Intraocular bleeding =< 6 months prior to randomization
  * Gastrointestinal bleeding and/or endoscopically proven ulcer =< 6 months prior to randomization
  * Head trauma or major trauma =< 1 month prior to randomization
  * Neurosurgery =< 2 weeks prior to randomization
  * Major surgery =< 1 week prior to randomization
  * Gross hematuria at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2025-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D McBane, Principal Investigator — Academic and Community Cancer Research United
Locations (32):
- United States (32):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin LAPS, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] McBane RD 2nd, Loprinzi CL, Zemla T, Tafur A, Sanfilippo K, Liu JJ, Garcia DA, Heun J, Gundabolu K, Onitilo AA, Perepu U, Drescher MR, Henkin S, Houghton D, Ashrani A, Billett H, McCue SA, Lee MK, Le-Rademacher JG, Wysokinski WE; EVE trial investigators. Extending venous thromboembolism secondary prevention with apixaban in cancer patients. The EVE trial. J Thromb Haemost. 2024 Jun;22(6):1704-1714. doi: 10.1016/j.jtha.2024.03.011. Epub 2024 Mar 25. PMID 38537780
- [Derived] McBane RD 2nd, Loprinzi CL, Ashrani A, Lenz CJ, Houghton D, Zemla T, Le-Rademacher JG, Wysokinski WE. Extending venous thromboembolism secondary prevention with apixaban in cancer patients: The EVE trial. Eur J Haematol. 2020 Feb;104(2):88-96. doi: 10.1111/ejh.13338. Epub 2019 Nov 11. PMID 31606897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 patients enrolled in arm 1 and 5 patients enrolled in arm 2 did not begin treatment and therefore are not included in the participant flow table.
Groups:
- Group I (2.5mg Dose Apixaban): Patients receive lower dose apixaban PO BID for 365 days. >
  > Apixaban: Given PO
- Group II (5mg Dose Apixaban): Patients receive higher dose apixaban PO BID for 365 days. >
  > Apixaban: Given PO
Period: Overall Study
Arm/Group | Group I (2.5mg Dose Apixaban) | Group II (5mg Dose Apixaban)
Started | 179 | 181
Completed | 111 | 109
Not Completed | 68 | 72
Not completed — Withdrawal by Subject | 11 | 15
Not completed — Adverse Event | 22 | 22
Not completed — Alternative Therapy | 0 | 3
Not completed — Other Complicating Disease | 9 | 5
Not completed — Death | 21 | 16
Not completed — Physician Decision | 2 | 2
Not completed — Disease Progression | 2 | 8
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group I (2.5mg Dose Apixaban): Patients receive lower dose apixaban PO BID for 365 days.>
  > Apixaban: Given PO
- Group II (5mg Dose Apixaban): Patients receive higher dose apixaban PO BID for 365 days.>
  > Apixaban: Given PO
- Total: Total of all reporting groups
Arm/Group | Group I (2.5mg Dose Apixaban) | Group II (5mg Dose Apixaban) | Total
Number analyzed (Participants) | 179 | 181 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (10.96) | 64.3 (10.72) | 64.0 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 107 | 199
  Male | 87 | 74 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 171 | 176 | 347
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 168 | 169 | 337
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 179 | 181 | 360
Primary Tumor Site [Count of Participants; unit: Participants]
  Brain/CNS | 3 | 5 | 8
  Breast | 10 | 25 | 35
  Colon/rectum/pancreas/stomach | 44 | 45 | 89
  ENT | 0 | 1 | 1
  Genitourinary | 0 | 3 | 3
  Gynecologic | 19 | 17 | 36
  Kidney/bladder | 8 | 9 | 17
  Liver/bile duct | 6 | 3 | 9
  Lung/bronchus | 26 | 17 | 43
  Lymphoma/Myeloma/Leukemia | 34 | 16 | 50
  Melanoma | 1 | 0 | 1
  Other | 4 | 3 | 7
  Prostate | 5 | 6 | 11
  Sarcoma | 5 | 4 | 9
  Skin | 1 | 3 | 4
  Thyroid | 2 | 3 | 5
  Tongue/mouth/pharynx | 0 | 2 | 2
  Upper Gastrointestinal | 3 | 2 | 5
  Uterine cervix/corpus | 8 | 17 | 25
ECOG Performance Status [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 97 | 96 | 193
    1 | 73 | 80 | 153
    2 | 9 | 5 | 14
Location of Initial Thrombosis [Count of Participants; unit: Participants]
  Deep-vein thrombosis (including atypical VTE) | 82 | 86 | 168
  Pulmonary embolism | 97 | 95 | 192

OUTCOME MEASURES:

1. Primary Outcome: CIF of Major or Clinically Relevant Non-major Bleeding Combined With Death as Competing Risk
Description: Incidence of major bleeding and clinically relevant non-major bleeding will be estimated using the cumulative incidence function (CIF) with death without major bleeding or clinically relevant non-major bleeding and with adverse events that results in termination of treatment (including vascular events) as competing risks. The time to event is defined as the time from randomization to the first occurrence of a major bleeding, a clinically relevant non-major bleeding, death without major bleeding or clinically relevant non-major bleeding, or an adverse event that results in termination of treatment. Patients who were lost to follow-up, who withdrew informed consent before the end of the predefined study duration will be censored at the last day the patient had a complete assessment for study outcomes within the intended study period. The difference in the incidences of the combined endpoint at 12 months between treatment arms will be estimated along with a 95% confidence interval
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group I (2.5mg Dose Apixaban) | Group II (5mg Dose Apixaban)
Number analyzed (Participants) | 179 | 181
proportion of participants | 9.6 [6.0 to 15.4] | 13.5 [9.1 to 20.0]
Statistical Analysis 1: Comparison: Group I (2.5mg Dose Apixaban) vs Group II (5mg Dose Apixaban); Test type: Superiority; p = 0.3117, Gray Test P-value; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.38 to 1.37]

2. Secondary Outcome: Proportion of Patients Who Experienced at Least One Bleeding Event
Description: Incidence of major bleeding and clinically relevant non-major bleeding will be estimated using the cumulative incidence function (CIF) with death without major bleeding or clinically relevant non-major bleeding and with adverse events that results in termination of treatment (including vascular events) as competing risks. The time to event is defined as the time from randomization to the first occurrence of a major bleeding, a clinically relevant non-major bleeding, death without major bleeding or clinically relevant non-major bleeding, or an adverse event that results in termination of treatment. Patients who were lost to follow-up, who withdrew informed consent before the end of the predefined study duration will be censored at the last day the patient had a complete assessment for study outcomes within the intended study period. The difference in the incidences of the combined endpoint at 6 months between treatment arms will be estimated along with a 95% confidence interval.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group I (2.5mg Dose Apixaban) | Group II (5mg Dose Apixaban)
Number analyzed (Participants) | 179 | 181
proportion of participants | 4.9 [2.5 to 9.7] | 5.8 [3.0 to 10.9]
Statistical Analysis 1: Comparison: Group I (2.5mg Dose Apixaban) vs Group II (5mg Dose Apixaban); Test type: Superiority; p = 0.9970, Gray Test P-value; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.40 to 2.53]

3. Secondary Outcome: Cumulative Incidence Function of DVT/PE Treating Death or AE Resulting in End of Treatment as Competing Risk by Study Arm
Description: For the secondary outcome analysis, the time from starting treatment to the first event of the composite deep vein thrombosis (DVT)/pulmonary embolism (PE) outcome will be analyzed using the same method described in the section for primary outcome plan. For this outcome, death without DVT/PE and adverse events leading to termination of treatment will be treated as the competing risks.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group I (2.5mg Dose Apixaban) | Group II (5mg Dose Apixaban)
Number analyzed (Participants) | 179 | 181
proportion of participants | 5.8 [3.2 to 10.6] | 7.1 [4.1 to 12.2]

ADVERSE EVENTS:
Time Frame: 29 months
Groups:
- Group I (2.5mg Dose Apixaban); Group II (5mg Dose Apixaban): Apixaban: Given PO
Arm/Group | Group I (2.5mg Dose Apixaban) | Group II (5mg Dose Apixaban)
All-Cause Mortality (participants affected / at risk) | 26/179 | 22/181
Serious Adverse Events (participants affected / at risk) | 70/179 | 69/181
Other Adverse Events (participants affected / at risk) | 93/179 | 75/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (2.5mg Dose Apixaban) (N=179) | Group II (5mg Dose Apixaban) (N=181)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 3 (3)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 4 (4)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 4 (4) | 3 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (7) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (3) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (6) | 6 (7)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (2)
Death NOS (General disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 3 (3) | 4 (4)
Fever (General disorders) | 1 (1) | 2 (2)
Gen disord and admin site conds-Oth spec (General disorders) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Sudden death NOS (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (3) | 2 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 (3) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 6 (7) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 6 (7) | 9 (11)
Skin infection (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urostomy stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (3) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (7) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 3 (3) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 (24) | 19 (19)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Muscle weakness right-sided (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Stroke (Nervous system disorders) | 2 (2) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 6 (7) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 2 (3) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 4 (4) | 4 (4)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I (2.5mg Dose Apixaban) (N=179) | Group II (5mg Dose Apixaban) (N=181)
Anemia (Blood and lymphatic system disorders) | 25 (53) | 23 (39)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 6 (8) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 2 (3)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 1 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 6 (9) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (2) | 4 (5)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Pancreatitis (Gastrointestinal disorders) | 1 (4) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 9 (10) | 2 (2)
Fatigue (General disorders) | 14 (26) | 4 (4)
Fever (General disorders) | 2 (2) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 3 (4) | 1 (1)
Localized edema (General disorders) | 1 (2) | 1 (1)
Neck edema (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 3 (4) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 4 (5) | 3 (4)
Lung infection (Infections and infestations) | 1 (1) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (3) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4) | 2 (2)
Alkaline phosphatase increased (Investigations) | 3 (20) | 7 (13)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 4 (4)
Blood bilirubin increased (Investigations) | 1 (2) | 2 (2)
Cardiac troponin T increased (Investigations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 5 (20) | 1 (2)
INR increased (Investigations) | 3 (3) | 1 (1)
Investigations - Other, specify (Investigations) | 2 (2) | 2 (2)
Lymphocyte count decreased (Investigations) | 18 (58) | 11 (14)
Neutrophil count decreased (Investigations) | 8 (13) | 6 (7)
Platelet count decreased (Investigations) | 12 (19) | 7 (14)
Urine output decreased (Investigations) | 1 (1) | 1 (1)
Weight loss (Investigations) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 10 (18) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (14) | 5 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (20) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 5 (6)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (4)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Dysgeusia (Nervous system disorders) | 1 (2) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 4 (8) | 3 (7)
Hematuria (Renal and urinary disorders) | 5 (5) | 8 (8)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (1) | 2 (2)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 12 (13) | 5 (5)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT03080883/Prot_SAP_ICF_000.pdf